CLINICAL TRIAL: NCT00754039
Title: The Effects of the Combination of Welchol and Tricor Compared to TriCor Alone in Patients With Mixed Hyperlipidemia
Brief Title: Study to Compare Welchol and TriCor to TriCor Alone in Patients With High Cholesterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Senior Director, Metabolic Medical Research, Daiichi Sankyo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WEL-403
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia; Hyperlipidemia, Familial Combined
Keywords: Mixed hyperlipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemia, Familial Combined; Hyperlipoproteinemia Type II | interventions — Colesevelam Hydrochloride; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Welchol + TriCor
  Interventions: Drug: colesevelam HCl tablets and fenofibrate tablets
- 2 (Placebo Comparator): Welchol + placebo
  Interventions: Drug: fenofibrate tablets and Welchol placebo tablets

INTERVENTIONS:
Drug: colesevelam HCl tablets and fenofibrate tablets — Colesevelam 625 mg tablets - 6 tablets/day Fenofibrate 160 mg tablet - 1/day
  Arms: 1
Drug: fenofibrate tablets and Welchol placebo tablets — fenofibrate tablets 160 mg - 1/day + Welchol placebo tablets - 6/day
  Arms: 2
Drug: fenofibrate tablets and Welchol placebo tablets — fenofibrate 160 mg tablet - 1/day and Welchol placebo tablets - 6/day
  Arms: 2

SUMMARY:
The primary objective of this study is to compare the effect of Welchol in combination with TriCor compared to TriCor alone on low-density lipoprotein cholesterol (LDL-C) in patients with high cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* 30-70 years of age
* History of mixed hyperlipidemia
* Prescribed a Step 1 diet at least 30 days prior to screening
* Women were not pregnant, breast-feeding, or plan to become pregnant during the study
* Women had a hysterectomy or tubal ligation, were post-menopausal, or practiced reliable birth control procedures
* Serum LDL-C >/= 115 mg/dL; Serum TG >/= 150 & < 750 mg/dL

Exclusion Criteria:

* BMI >40
* HbA1C > 10%
* Type 1 diabetes
* Intolerance to fibrates
* History of intolerance to colesevelam HCl
* History of swallowing disorders or intestinal motility disorders
* Any other disorder that might interfere with the conduct of the study
* History of drug or alcohol abuse
* Recent (within 28 days) history of cardiac disease (MI, CHF, CABG, etc.)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2003-02; Primary Completion 2003-09 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
% change in LDL-C from baseline | 6 weeks

SECONDARY OUTCOMES:
The absolute change in LDL-C from baseline | 6 weeks
The absolute change and % change in LDL-C from week -8 (untreated) | 14 weeks
The percentage of patients who achieved target LDL-C | 6 Weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Longwood, Florida
  - Ocala, Florida
  - Winterpark, Florida
  - Chicago, Illinois
  - Lombard, Illinois
  - Overland Park, Kansas
  - Stateville, North Carolina
  - Cincinnati, Ohio
  - San Antonio, Texas
  - Richmond, Virginia